CLINICAL TRIAL: NCT04835207
Title: Metabolic Profile as a Predictor of No-reflow in Diabetic Patients Treated With Primary Percutaneous Coronary Intervention ( PCI ) .
Brief Title: Metabolic Profile as a Predictor of No-reflow in Diabetic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: El Zahraa Gamal (Other)
Responsible Party: Sponsor-Investigator, El Zahraa Gamal, Metabolic profile as a predictor of no reflow in diabetic patients treated with primary Percutaneous Coronary Intervention (PCI) ., Assiut University
Organization: Assiut University (Other)
Other Study IDs: primary ( PCI )
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Acute Myocardial Infarction (AMI)
MeSH Terms: interventions — Cholesterol, LDL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 1- LDL-C (low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotein cholesterol) Ratio. 2- Glycemia will be assessed : RBS ( random blood sugar ) . 3- S — Blood samples were obtained before PCI, and the following parameters will be measured: 1- LDL-C (low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotein cholesterol) Ratio. 2- Glycemia will be assessed : RBS ( random blood sugar ) . 3- S

SUMMARY:
to find metabolic factors that correlate with the development of no-reflow phenomenon that may help prevent its occurrence

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) with its accompanying adverse sequelae is one of the most common causes of morbidity and mortality in the world .

Although reperfusion techniques for ST- elevation myocardial infarction (STEMI ) are constantly improving, no-reflow can still lead to poor prognosis .

At present, the exact mechanism of no-reflow remains unclear, but clinical and laboratory findings suggest that it is related to the embolism of the capillary bed, ischemic injury, vascular endothelial dysfunction, production of oxygen free radical , and other factors .

The no-reflow phenomenon is one of complications of poor functional and clinical outcomes for patients with (AMI) .

The no-reflow phenomenon is present in 25% to 30% of patients with (AMI) underwent successful coronary recanalization, as shown by angiography . The myocardial no-reflow phenomenon is associated with a reducution of antegrade myocardial blood flow inspite of an open infarct-related artery in patients with (STEMI ) undergoing (PCI) . Importantly, no-reflow is known to be related to unfavorable clinical outcome and prognosis . The cause of this complex phenomenon is the variable combination of four pathogenetic components: distal atherothrombotic embolization, ischemic injury, reperfusion injury and susceptibility of coronary microcirculation to injury . As a consequence, appropriate strategies are expected to prevent or treat these components are expected to avoid the no-reflow. Coronary reperfusion therapy is widely performed in patients with (AMI) . However, in spite of patency of the infarct-related artery , there is no guarantee of salvage of myocardium at risk of ischemia .The no-reflow phenomenon is found in >30% of patients after thrombolysis or catheter-based (PCI) for (AMI) . It is important, therefore, to be able to predict which lesions are high risk for no reflow before beginning PCI .

Many of the well-accepted risk factors for no-reflow are similar to other well-accepted cardiovascular risk factors, such as hypertension, smoking, dyslipidemia, diabetes, and other inflammatory processes. As such, there are some generally accepted measures associated with a lower incidence of no-reflow following PCI for STEMI. For example, in patients with diabetes, optimal blood sugar control before the procedure can reduce the occurrence of no-reflow .

There are numerous recognized risk factors for the development of coronary artery disease (CAD), one of the best known is the association between blood lipids and CAD . Several prospective studies have established that the risk of cardiac morbidity and mortality is directly related to the concentration of plasma cholesterol. ' The most prevalent view is that the increased risk of myocardial infarction associated with elevated plasma cholesterol levels can be adequately explained on the basis of the increase in number and severity of coronary atherosclerotic vascular lesions . .

Hyperglycemia is associated with The increased mortality in patients with acute myocardial infarction which caused by a larger infarct size, a high incidence of congestive heart failure, and cardiogenic shock, and death after AMI., . However, the underlying mechanisms of these deleterious effects of hyperglycemia are not well understood Uric acid (UA) is a byproduct the terminal steps of purine catabolism, . uric acid synthesis is increased under tissue ischemia. Therefore, elevated uric acid may affect prognosis of (AMI). A few studies have doucomented that UA is associated with therapeutic results in patients with AMI. UA level is appeared to be related to infarct size and hemodynamic derangement. Although prompt restoration of myocardial blood flow is very important for patients with AMI, high levels of UA are doucoumented to be significantly associated with the presence of slow coronary flow

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with ST- elevation myocardial infarction (STEMI ) treated with primary Percutaneous Coronary Intervention ( PCI ) .

Exclusion Criteria:

diabetic patients with ST- elevation myocardial infarction (STEMI ) treated with primary Percutaneous Coronary Intervention ( PCI ) : but have

* (1) a history of an unprotected left main artery with severe liver and kidney diseases or coronary artery bypass grafting .

  (2) patients who had valvular disease or cardiomyopathy . (3) severe dissection, thromboembolism in other parts, or vasospasm; and known malignancy .

  (4) patients with contraindications for anticoagulant therapy, such as active visceral hemorrhage, hemorrhagic stroke, or ischemic stroke within half a year (including transient ischemic attack), or aortic dissection, or patients with hematological diseases complicated with coagulation disorders .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: diabetic patients with STEMI treated with primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
detection correlation between DM and no-reflow phenomenon | baseline
  measurment of random blood sugar in diabetic patients treated with primary Percutaneous Coronary Intervention ( PCI ) .and show its effects on reflow

SECONDARY OUTCOMES:
detection correlation between other metabolic factors as serum uric acid and no-reflow phenomenon | baseline
  Blood samples were obtained before PCI, and the following parameters will be measured :Serum Uric acid : S .UA
detection correlation between other metabolic factors as LDL\HDL and no-reflow phenomenon | baseline
  Blood samples were obtained before PCI, and the following parameters will be measured :(LDL\HDL :(low-density lipoprotein cholesterol)| and HDL-C(high-density lipoprotei

REFERENCES:
- [Background] Bernstein JM, Lee J, Conboy K, Ellis E, Li P. The role of IgE mediated hypersensitivity in recurrent otitis media with effusion. Am J Otol. 1983 Jul;5(1):66-9. No abstract available. PMID 6683937